CLINICAL TRIAL: NCT03063437
Title: Phase II Randomized, Double Blind, Placebo-controlled, Parallel Group Trial of Encapsulated Fecal Microbiota Transplantation for Vancomycin Resistant Enterococcus Decolonization
Brief Title: A Trial of Encapsulated Fecal Microbiota for Vancomycin Resistant Enterococcus Decolonization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Microbiome Health Research Institute (Other)
Collaborators: University of Wisconsin, Madison (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200-2016-91948
Record Dates: First submitted 2017-02-17; First posted 2017-02-24 (Actual); Results first posted 2020-02-05 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Antibiotic Resistant Strain
Keywords: vancomycin resistant enterococcus; VRE; decolonization; VRE colonization; fecal microbiota transplantation; FMT; FMT capsule; capsule; antimicrobial resistance; antibiotic resistance; MDRO; multidrug-resistant organism; OpenBiome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active: Encapsulated Fecal Microbiota Preparation (Experimental): Single dose of oral, encapsulated fecal microbiota preparation (30 capsules per dose) with follow-up at 3 days, 10 days, 28 days, and 6 months.
  Interventions: Biological: Encapsulated fecal microbiota preparation
- Placebo: Encapsulated Placebo (Placebo Comparator): Single dose of oral, placebo capsule (30 capsules per dose) with follow-up at 3 days, 10 days, and 28 days, and 6 months.
  Interventions: Biological: Encapsulated placebo

INTERVENTIONS:
Biological: Encapsulated fecal microbiota preparation — 30 capsules
  Arms: Active: Encapsulated Fecal Microbiota Preparation
Biological: Encapsulated placebo — 30 capsules
  Arms: Placebo: Encapsulated Placebo

SUMMARY:
The objective of this study is to provide preliminary insight into the safety and efficacy of fecal microbiota transplantation (FMT) for the eradication of gastrointestinal carriage of vancomycin-resistant Enterococcus.

DETAILED DESCRIPTION:
Note: The Protocol and Statistical Analysis Plan document contains modifications from what is on file at the FDA to reflect redactions and formatting requirements for public posting on ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older at the time of enrollment.
* Able to provide signed and dated informed consent.
* Identified as VRE-positive by a stool culture within last 14 days.
* Women of childbearing potential in sexual relationships with men must use an acceptable method of contraception§ from 30 days prior to enrollment until 4 weeks after completing study treatment.
* Males must agree to avoid impregnation of women during and for four weeks after completing study treatment through use of an acceptable method of contraception*.

  * Includes, but is not limited to, barrier with additional spermicidal foam or jelly, intrauterine device, hormonal contraception (started at least 30 days prior to study enrollment), intercourse with men who underwent vasectomy.

    * Includes, but is not limited to, barrier with additional spermicidal foam or jelly and vasectomy.

Exclusion Criteria:

* Female patient who are pregnant, lactating or planning on becoming pregnant during study. Female patients of childbearing potential will undergo a pregnancy test, and be excluded from the study if positive.
* Inability (e.g. dysphagia) to or unwilling to swallow capsules.
* Active antibiotic resistant bacteria (ARB) or gastrointestinal infection at time of enrollment.
* Patient received antibiotics in the last 48 hours. Patients will be eligible to enroll if antibiotic therapy is discontinued for at minimum 48 hours prior to randomization. Does not include antibiotics used for prophylaxis or topical antibiotics.
* Requires continued antibiotic use or anticipates antibiotic use in the upcoming 4 weeks. Does not include antibiotics used for prophylaxis or topical antibiotics.
* Unwilling to withhold probiotics for a minimum of 48 hours prior to providing a screening stool sample.
* Known or suspected toxic megacolon and/or known small bowel ileus.
* Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment. This does not include appendectomy or cholecystectomy.
* History of total colectomy or bariatric surgery.
* Admitted to or expected to an intensive care unit for medical reasons (not just boarding). Patients residing in a nursing home, long-term care facility or rehabilitation center may be enrolled.
* Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for active malignancy. Patients on maintenance chemotherapy may be enrolled only after consultation with medical monitor.
* Unable or unwilling to comply with protocol requirements.
* Expected life expectancy < 6 months
* Previous FMT or microbiome-based products at any time excluding this study.
* Patients with a history of severe anaphylactic or anaphylactoid food allergy.
* Solid organ transplant recipients ≤ 90 days post-transplant or on active treatment for rejection.
* Neutropenia (≤500 neutrophils/mL) or other severe immunosuppression. Anti-TNF will be permitted. Patients on monoclonal antibodies to B and T cells. glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine, methotrexate), calcineurin inhibitors (tacrolimus, cyclosporine) and mycophenolate mofetil may be enrolled only after consultation with the medical monitor.
* If at risk for CMV/EBV associated disease (at investigator's discretion, e.g. immunocompromised), negative IgG testing for cytomegalovirus (CMV) or Epstein Barr Virus (EBV).
* A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2019-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Majdi Osman, MD, MPH, Principal Investigator — Microbiome Health Research Institute d/b/a OpenBiome
Locations (2):
- United States (2):
  - IU Health University Hospital, Indianapolis, Indiana
  - University of Wisconsin University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the listed tertiary academic hospitals from August 15, 2017 to September 30, 2018.
Groups:
- Placebo: Encapsulated Placebo: Single dose of oral, placebo capsule (30 capsules per dose) with follow-up at 3 days, 10 days, 28 days, and 6 months.
Period: Overall Study
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With VRE Decolonization
Description: VRE decolonization is defined by absence of VRE on stool culture using standard clinical laboratory techniques at Day 10 (± 3 days) after randomization.
Time Frame: Day 10 (±3 days) after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 4 | 5
Participants | 1 | 1

2. Primary Outcome: Percentage of Participants With an Adverse Event (AE); Severe Adverse Event (SAE); and Newly Acquired Transmissible Infectious Diseases Which Are Considered Adverse Events of Special Interest (AESI)
Description: Percentage of participants with an adverse event (AE); severe adverse event (SAE); and newly acquired transmissible infectious diseases which are considered adverse events of special interest (AESI) through Day 10 (± 3 days) after randomization.
Time Frame: Day 10 (±3 days) after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 4 | 5
Participants | 3 | 5

3. Secondary Outcome: Percentage of Participants With VRE Infection
Description: Percentage of participants with VRE infection, defined as an associated bacteremia, urinary tract infection, or wound-related infection.
Time Frame: Week 4 (±5 days) after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

4. Secondary Outcome: Percentage of Participants With ARB Colonization on Day 10 Following Fecal Microbiota Transplantation (FMT)
Description: Percentage of participants with other antibiotic resistant bacteria (ARB) colonization
Time Frame: Day 10 (± 3 days) after randomization
Population: Data not collected as no participants in the trial entered the study colonized with an ARB other than VRE
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Participants With ARB Infection 4 Weeks Following FMT
Description: Percentage of participants with composite ARB infection
Time Frame: Week 4 (±5 days) after randomization
Population: Data not collected as no participants in the trial entered the study colonized with an ARB other than VRE
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Days Between FMT and VRE Colonization and Infection Occurs
Description: Time (in days) from randomization until the study day when VRE colonization and infection occurs
Time Frame: Up to 6 months after randomization
Population: Data not collected as no participants in the trial were colonized and infected by VRE following randomization.
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: VRE Decolonization Among Immunocompromised Patients
Description: Percentage of participants with VRE decolonization among immunocompromised patients
Time Frame: Day 10 (± 3 days) after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 4 | 4
Participants | 1 | 1

8. Secondary Outcome: Adverse Events Within 4 Weeks Following FMT
Description: Percentage of participants with an adverse event (AE)
Time Frame: Week 4 (±5 days) after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 4 | 5
Participants | 3 | 5

9. Secondary Outcome: Serious Adverse Events Within 4 Weeks Following FMT
Description: Percentage of participants with a serious adverse event (SAE)
Time Frame: Week 4 (±5 days) after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

10. Secondary Outcome: Newly Acquired Transmissible Infectious Diseases Which Are Considered Adverse Events of Special Interest (AESI)
Description: Percentage of participants with newly acquired transmissible infectious diseases which are considered adverse events of special interest (AESI)
Time Frame: Week 4 (±5 days) after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 4 | 5
Participants | 0 | 0

11. Secondary Outcome: Serious Adverse Events Within 6 Months Following FMT
Description: Percentage of participants with a Serious Adverse Event (SAE)
Time Frame: Month 6 (±14 days) phone safety assessment after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
Number analyzed (Participants) | 4 | 5
Participants | 2 | 1

12. Other Pre Specified Outcome: Microbiome Disruption
Description: To evaluate the microbiome disruption index (MDI) by 16s rRNA sequencing): MDI-community and MDI-species
Time Frame: Day 3, day 10, week 4 after randomization.
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Engraftment Dynamics
Description: To evaluate the trends in VRE type/strain-level engraftment using whole genome sequencing among those colonized
Time Frame: 6 months following FMT
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 6 months after randomization,
Arm/Group | Active: Encapsulated Fecal Microbiota Preparation | Placebo: Encapsulated Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/5
Other Adverse Events (participants affected / at risk) | 3/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active: Encapsulated Fecal Microbiota Preparation (N=4) | Placebo: Encapsulated Placebo (N=5)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active: Encapsulated Fecal Microbiota Preparation (N=4) | Placebo: Encapsulated Placebo (N=5)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal distention (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Discolored stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) — General disorders and administration site conditions
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Throat pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Loss of appetite (General disorders) | 0 (0) | 1 (1)
Elevated liver function tests (Hepatobiliary disorders) | 1 (1) | 1 (1)
Polymyalgia rheumatica (Immune system disorders) | 0 (0) | 1 (1)
CMV re-activation (Infections and infestations) | 0 (0) | 1 (1) — Cytomegalovirus (CMV) re-activation
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/37/NCT03063437/Prot_SAP_000.pdf